CLINICAL TRIAL: NCT04024878
Title: NeoVax With Nivolumab in Patients With Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Ott, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-318
Record Dates: First submitted 2019-05-24; First posted 2019-07-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Nivolumab; Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stanfard Platinum (Experimental): * A total of 5 NeoVax immunizations will be administered over a 3-week period
  * Two booster vaccinations will be given at Week 12
  * Nivolumab administered by intravenous (IV) infusion over 30 minutes every 2 weeks.
  Interventions: Drug: Nivolumab; Biological: NeoVax
- Stanfard Platinum with Surgical or Core Needle Biopsy (Experimental): * A total of 5 NeoVax immunizations will be administered over a 3-week period
  * Two booster vaccinations will be given at Week 12
  * Nivolumab administered by intravenous (IV) infusion over 30 minutes every 2 weeks.
  * Will undergo required surgical or core needle biopsy at first recurrence with progression free interval
  Interventions: Drug: Nivolumab; Biological: NeoVax; Procedure: Core Needle Biopsy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (Opdivo®) is an antibody. An antibody is a common type of protein produced by the body that the immune system uses to find and destroy foreign molecules.
  Other Names: Opdivo
Biological: NeoVax — The vaccine will consist of up to 20 peptides as well as a drug that activates the immune system called Poly-ICLC. Poly-ICLC (also called Hiltonol) is an experimental "viral mimic" and an activator of immunity
Procedure: Core Needle Biopsy — Surgical procedure
  Arms: Stanfard Platinum with Surgical or Core Needle Biopsy

SUMMARY:
This research study is evaluating a new type of vaccine called "Personalized NeoAntigen Cancer Vaccine" in combination with Nivolumab (Opdivo®) for ovarian cancer.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational Personalized Cancer Vaccine in combination with Nivolumab (Opdivo®). "Investigational" means that the Personalized Cancer Vaccine is being studied. It also means that the U.S. Food and Drug Administration (FDA) has not approved the Personalized Cancer Vaccine as a treatment for any disease.

The U.S. Food and Drug Administration (FDA) has not approved Nivolumab for this specific disease but it has been approved for other uses.

The purpose of this study is to determine if it is possible to make and administer safely a vaccine against ovarian cancer by using information gained from specific characteristics of the participant's own ovarian cancer. It is known that ovarian cancers have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the body fight tumor ovarian cancer cells. The study will examine the safety of the vaccine when given at several different time points and will examine the blood cells for signs that the vaccine induced an immune response.

Ovarian cancer cells will be obtained from the tumor through a biopsy. The genetic material contained in the ovarian cancer cells will be examined for the presence of tumor-specific mutations. This information will be used to prepare small protein fragments, which are called "peptides". The vaccine will consist of up to 20 of these peptides as well as a drug that activates the immune system called Poly-ICLC.

Poly-ICLC (also called Hiltonol) is an experimental "viral mimic" and an activator of immunity. Poly-ICLC binds proteins on the surface of certain immune cells to make it appear as if a virus is present. When the cells detect the vaccine, they think it is a virus and turn on the immune system. Poly-ICLC is a compound that has been used to help the body in its fight against cancer. Poly-ICLC will be mixed with NeoAntigen peptides and administered as an injection given underneath the skin. Poly-ICLC is an investigational drug, meaning the FDA has not approved it as a treatment for any disease.

Nivolumab (Opdivo®) is an antibody that has been approved by the United States Food and Drug Administration (FDA) for the treatment of metastasic lung cancer, metastasic melanoma, advanced renal cell carcinoma, recurrent or metastasic carcinoma of the neck, hepatocellular carcinoma, advanced or metastasic urothelial carcinoma, metastasic colorectal cancer, and relapsed or progressed Hodgkin Lymphoma.

An antibody is a common type of protein produced by your body that the immune system (a system that defends the body against potentially harmful particles) uses to find and destroy foreign molecules (particles not typically found in the body) such as bacteria and viruses. Antibodies can also be produced in the laboratory for use in treating patients. There are now several approved antibodies for the therapy of cancer and other diseases.

Nivolumab is an antibody that acts against PD-1. PD-1 is a molecule that controls a part of the immune system by shutting it down. Researchers believe that one way cancers can escape the immune system could also be by blocking it out so. An antibody against PD-1 can stop PD-1 from turning off the immune system, allowing the immune reaction to continue. The body's immune reaction may help the body to destroy cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial ovarian cancer, primary peritoneal or fallopian tube cancer. High grade serous, high grade endometrioid, clear cell and carcinosarcoma (carcinosarcomas only with high grade serous epithelial component) histologies are allowed. Low grade histologies and mucinous histology are not allowed.
* Participants must be classified into one of two cohorts:
* Cohort A: Patients with newly diagnosed stage IIIC or stage IV epithelial ovarian, fallopian tube, or primary peritoneal cancer who are planned to undergo neoadjuvant chemotherapy. Patients must be candidates for platinum-based chemotherapy and previously untreated. At the time of pre-screening consent, patients must have disease that is amenable to biopsy and are agreeable and can safely undergo biopsy.
* Cohort B: Patients with recurrent (first recurrence only) epithelial ovarian, primary peritoneal or fallopian tube cancer with platinum sensitive disease defined as disease progression greater or equal than 6 months but not more than 18 months after completion of their last dose of first line platinum chemotherapy. Prior hormonal therapy is allowed but no other therapy for recurrence is allowed, including no chemotherapy, no targeted therapy, and no antiangiogenic therapy. Maintenance therapy after first line chemotherapy is allowed. At the time of pre-screening consent, patients must have measurable disease by RECIST 1.1 and disease that is amenable to biopsy and are agreeable and can safely undergo biopsy.
* Eastern Cooperative Group (ECOG) performance status ≤2 (please see Appendix A)
* Age ≥18 years
* Patients must have adequate organ and bone marrow function:

  * Haemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * White blood cells (WBC) > 2x109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
* Negative serum β-HCG or urine pregnancy test
* Ability to understand and the willingness to sign a written informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment with Nivolumab and 5 months after the last dose of study treatment {i.e., 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives}.

Patients of non-childbearing potential are defined as those fulfilling at least one of the following criteria:

* Have undergone a documented hysterectomy and/or bilateral oophorectomy;
* Have medically confirmed ovarian failure; or
* Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state

Exclusion Criteria:

* Non-epithelial tumors or ovarian tumors with low malignant potential (i.e. borderline tumors)
* Mucinous or low grade histologies (i.e. low grade serous or low grade endometrioid)
* Cohort A and B patients who have signed prescreening consent form and then, in the opinion of the investigator, have progressed after 3 or 4 cycles of platinum-based chemotherapy, are ineligible for the treatment part of the study and no vaccine will be manufactured
* Prior immunotherapy with IL-2, IFN-α, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte associated antigen 4 (anti-CTLA-4) antibody (including Ipilimumab), or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Major surgery (other than debulking surgery for ovarian, primary peritoneal or fallopian tube cancer) for any reason within 4 weeks prior to initiation of vaccination and/or incomplete recovery from surgery
* Known brain metastases or leptomeningeal metastases because of their poor prognosis and because patients often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. A scan to confirm the absence of brain metastases is not required.
* Active or history of autoimmune disease (known or suspected). Exceptions are permitted for vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring only hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to the first dose of study drug (Nivolumab). Inhaled or topical steroids and adrenal replacement doses (≤ 10 mg daily prednisone equivalents) are permitted in the absence of active autoimmune disease.
* Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illnesses unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, interfere with participation in this study.
* Known allergy to tetanus toxoid
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
* Pregnant women are excluded from this study because Nivolumab, personalized neoantigen peptides, and Poly-ICLC are agents with unknown risks to the developing fetus.
* Nursing women are excluded from this study because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with Nivolumab, personalized neoantigen peptides, and Poly-ICLC.
* Have a history of an invasive malignancy, except for the following circumstance: individuals with a history of invasive malignancy are eligible if they have been disease-free for at least 2 years or are deemed by the investigator to be at low risk for recurrence of that malignancy; individuals with the following cancers are eligible if diagnosed and treated carcinoma in situ of the breast, oral cavity or cervix, localized prostate cancer, basal cell or squamous cell carcinoma of the skin.
* Participants who are receiving any other investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients pre-srceened who have enough neoantigens for generation of the vaccine, are not platinum refractory, and who initiate vaccination | 2 years
  To demonstrate that regimen of NeoVax with Nivolumab is feasible and safe for the treatment of patients with ovarian cancer.
Overall incidence of treatment-emergent AEs, SAEs, AEs of at least Grade 3 severity, related AEs, and AEs leading to withdrawal of treatment will be described | 2 years
  Safety analysis will be performed on all patients who receive at least one dose of the NeoVax.
The rates of autoimmune effects | 2 years

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
Duration of Response | 2 years
Progression Free Survival | 2 Years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation